CLINICAL TRIAL: NCT00926211
Title: Safety and Efficacy of Computer-Assisted vs. Manual Hair Follicle Harvest: A Comparative Hair Count Study
Brief Title: Computer-Assisted Versus Manual Hair Harvest Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Restoration Robotics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RR-09-0002
Record Dates: First submitted 2009-06-19; First posted 2009-06-23 (Estimated); Results first posted 2011-12-08 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2011-09

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computer-Assisted (Experimental): Hair harvest using the computer-assisted system
  Interventions: Device: ARTAS™ System
- Manual Harvest (Active Comparator): Hair harvesting via manual technique
  Interventions: Procedure: Manual Hair Harvest

INTERVENTIONS:
Device: ARTAS™ System — Hair harvest using a computer-assisted system
  Arms: Computer-Assisted
Procedure: Manual Hair Harvest — Hair harvesting via the manual technique
  Arms: Manual Harvest

SUMMARY:
The objective of this clinical study is to investigate and compare the safety and efficacy of the Restoration Robotics Computer-Assisted Harvesting System to the manual hair follicle harvesting method following a nine-month period of post-procedural evaluation.

DETAILED DESCRIPTION:
A major technical step in hair transplantation is harvesting of the hair follicles. There are two accepted techniques for obtaining the hair grafts that are transplanted during the procedure. The first is donor strip harvest and stereomicroscopic dissection of the follicular unit grafts. The second is dissection and extraction of the follicular unit graft directly from the patient's scalp referred to as Follicular Unit Extraction or "FUE". Potential benefits of the FUE technique may be less scalp scarring in the Donor Area, less patient discomfort and faster wound healing. Although the FUE approach to harvest has highly desirable attributes, it is technically difficult to perform, labor intensive, tedious and requires an excessive amount of time to harvest follicular units. These procedural factors have prevented the FUE approach from gaining wider adoption.

Restoration Robotics, Inc. has developed the Restoration Robotics ARTAS™ Computer-Assisted Harvesting System to assist physicians in the harvest of hair follicles during hair transplantation procedures. The System mimics the manual FUE approach to harvesting follicular units and has the potential to solve the technical challenges inherent in the manual FUE technique. The ARTAS™ System is capable of identifying and harvesting hair follicles directly from the patient's scalp through a semi-automated process. The goal of the ARTAS™ System is to harvest the hair follicles while maintaining their critical anatomic structures intact.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male with clinical diagnosis of androgenic alopecia with Norwood-Hamilton grade of IV-VII
* Subject is 30 to 59 years old
* Subject has black or brown hair color
* Subject has straight hair
* Subject agrees to cut hair short (< 1 mm) on the scalp in the designated study areas for harvesting and implantation
* Subject agrees to have two dot tattoos placed on scalp
* Subject is able to understand and provide written consent; and
* Subject consents to post-operative follow-up per protocol.

Exclusion Criteria:

* Subject has preponderance of grey/white hair
* Subject has blonde hair
* Subject has red hair
* Subject uses hair dye
* Subject has prior history of hair restoration procedure(s) using the strip excision technique
* Subject has prior history of scalp reduction surgery(s)
* Subject has helical hair (curly hair)
* Subject has wavy hair
* Subject has bleeding diathesis
* Subject has active use of anti-coagulation medication
* Subject has used finasteride in the previous 6 months, or plans to use finasteride during the study
* Subject has used minoxidil in the previous 2 weeks, or plans to use minoxidil during the study; or
* Subject has any other condition that, in the opinion of the investigator, makes the subject inappropriate to take part in this study.

Ages: 30 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Canales, M.D., Study Director — Restoration Robotics
Locations (2):
- United States (2):
  - Berman Skin Institute, Palo Alto, California
  - A Practice of Hair Restoration, Walnut Creek, California

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from June 19, 2009 to September 23, 2010 at hair restoration clinics.
Pre-assignment Details: Once enrolled, subjects were scheduled for the treatment procedure. Subjects were randomized at the time of the treatment procedure.
Groups:
- Computer-Assisted and Manual Harvest: Each subject has a region of their scalp randomly assigned to be harvested by each method, the computer-assisted system or manual.
Period: Overall Study
Arm/Group | Computer-Assisted and Manual Harvest
Started | 36 (One additional subject was not randomized and did not receive the treatment procedure.)
Completed | 35
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Computer-Assisted and Manual Harvest
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 48.6 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 36
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Increase in Hair Follicles Present
Description: The increase in the number of hair follicles present at follow-up in each region compared to the number present at baseline.
Time Frame: Change from Baseline at 9 Months
Population: The analysis was based on intention to treat (ITT). Imputation technique was based LOCF.
Measure: Mean (Standard Deviation); unit: Hair follicles
Groups:
- Manual Harvest: Region of scalp with implanted follicles that were manually harvested.
- Computer-Assisted Harvest: Region of scalp with implanted follicles that were harvested using a computer-assisted system.
Arm/Group | Manual Harvest | Computer-Assisted Harvest
Number analyzed (Participants) | 36 | 36
Hair follicles | 16.9 (18.3) | 18.3 (18.0)
Statistical Analysis 1: Comparison: Manual Harvest vs Computer-Assisted Harvest; The hypothesis to be tested is one of non-inferiority. Tests of non-inferiority are one-sided tests and the significance level will be 0.025; Test type: Non-Inferiority or Equivalence — Initial planned sample size of 26 would provide approximately 90% power if the survival rate in the implanted transected follicles is at least 40%. Sample size used was 36 with 35 participants completing the 9 month study; p = 0.023, t-test, 1 sided — t-test comparison to the upper limit of the non-inferiority margin; Paired t-test compared to the non-inferiority margin of 4 follicles; Mean Difference (Net) = -1.4, 97.5% CI 1-sided [upper limit 3.9], Standard Deviation 15.5 — The number of implanted hairs surviving that were harvested using the computer assisted method was subtracted from the number of implanted hairs surviving that were harvested manually

2. Secondary Outcome: Proportion of Harvested Follicles Transected
Description: The proportion of harvested hair follicles that were transected by each harvest method.
Time Frame: Time of harvest (Baseline)
Measure: Mean (Standard Deviation); unit: Proportion of transected follicles
Arm/Group | Manual Harvest | Computer-Assisted Harvest
Number analyzed (Participants) | 36 | 35
Proportion of transected follicles | .264 (.112) | .219 (.146)
Statistical Analysis 1: Comparison: Manual Harvest vs Computer-Assisted Harvest; Paired data with each subject as their own control (treatment was randomly assigned to the left or right side of the scalp). Paired difference was analyzed; Test type: Non-Inferiority or Equivalence — Study was powered for the primary efficacy outcome; p < 0.001, t-test, 1 sided; Paired t-test; Mean Difference (Final Values) = .045, 97.5% CI 1-sided [lower limit -.004], Standard Deviation 0.146

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Computer-Assisted and Manual Harvest
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No